CLINICAL TRIAL: NCT00126620
Title: A Phase I Study of BAY 43-9006 (Sorafenib) in Combination With OSI-774 (Erlotinib; Tarceva) in Advanced Solid Tumors
Brief Title: Sorafenib and Erlotinib in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-042; CDR0000437855 (Registry Identifier: PDQ (Physician Data Query)); NCI-7178
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Erlotinib Hydrochloride; Sorafenib

ARMS (1):
- OSI-774 erlotinib) and Bay 43-9006 (Sorafenib) (Experimental): Sorafenib administered alone for a 1-week run-in period, and then both drugs e given together continuously, with every 28 days considered as a cycle. Three dose levels assessed.
  Interventions: Drug: erlotinib hydrochloride; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib and erlotinib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of sorafenib and erlotinib in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of sorafenib and erlotinib in patients with metastatic or unresectable solid tumors.

Secondary

* Determine the optimal biologically effective dose of this regimen that will lead to hypophosphorylation of epidermal growth factor receptor (EGFR), ERK, Akt, and vascular endothelial growth factor receptor (VEGFR), and inhibition of angiogenesis and apoptosis with tolerable toxicity in these patients.
* Correlate the pharmacokinetic profiles of this regimen with toxicity and biological activity in these patients.
* Determine, preliminarily, the antitumor activity of this regimen in these patients.
* Correlate phosphorylation status of EGFR, ERK, Akt, and VEGFR with antitumor activity of this regimen in these patients.

OUTLINE: This is a multicenter, open label, non-randomized, dose-escalation study.

Patients receive oral sorafenib alone once or twice daily on days -6 to 0*. Patients then receive oral sorafenib once or twice daily and oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Not considered part of course 1; considered a "run-in" period only.

Cohorts of 3-6 patients receive escalating doses of sorafenib and erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 10 patients are treated at the MTD.

After completion of study treatment, patients are followed at 4 weeks and then at least annually thereafter.

PROJECTED ACCRUAL: A total of 16-28 patients will be accrued for this study within 5-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Metastatic or unresectable disease
* Standard curative or palliative measures do not exist OR are no longer effective
* Measurable disease by radiography (for patients treated at the maximum tolerated dose [MTD] only)
* Tumor accessible for serial biopsies (for patients treated at the MTD only)
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No bleeding diathesis or coagulopathy

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times ULN
* PT INR ≤ 1.5 unless on full-dose warfarin

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 140 mm Hg or diastolic BP > 90 mm Hg despite medication)
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Ophthalmic

* No abnormalities of the cornea, including any of the following:

  * Dry eye syndrome
  * Sjögren's syndrome
  * Congenital abnormalities (e.g., Fuch's dystrophy)
  * Abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
  * Abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)

Gastrointestinal

* No active peptic ulcer disease that would impair the ability to swallow pills
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to undergo serial biopsies, positron emission tomography, and CT scanning (for patients treated at the MTD only)
* No ongoing or active infection
* No significant traumatic injury within the past 3 weeks
* No history of allergic reaction to drugs of similar chemical or biological composition to study drugs
* No psychiatric illness or social situation that would preclude study compliance
* No other condition that would impair the ability to swallow pills
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic hematopoietic colony-stimulating factors

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy (except for low dose, non-myelosuppressive radiotherapy) and recovered

Surgery

* More than 3 weeks since prior major surgery
* No prior surgical procedure affecting absorption

Other

* No prior sorafenib or erlotinib
* No other prior agents targeting Raf, vascular endothelial growth factor (VEGF), VEGF receptor, or epidermal growth factor receptor
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent CYP3A4 inducers (e.g., rifampin or Hypericum perforatum [St. John's wort])
* No other concurrent anticancer therapy
* Concurrent prophylactic anticoagulation therapy (e.g., low-dose warfarin) allowed provided PT INR < 1.1 times upper limit of normal (ULN)
* Concurrent full-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 allowed provided both of the following criteria are met:

  * Patient has an in range INR (between 2-3) while on a stable-dose of oral anti-coagulant OR a stable-dose of low molecular weight heparin
  * No active bleeding OR pathological condition that would confer a high risk of bleeding (e.g., tumor involving a major vessel or known varices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-09; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose | 28 days

SECONDARY OUTCOMES:
Pharmacodynamic outcomes | Pre study and cycle 1
Pharmacokinetic outcomes | Pre-study, cycle 1 and cycle 2
Antitumor activity | Every 8 wks
Correlation of EGFR, AKT, ERK and VEGFR with antitumor activity | If responses or prolonged stable disease are observed
EGFR activating mutations, gene amplification status, EGFR intron 1 polymorphism if responses or prolonged disease stabilization are seen | If responses or prolonged stable disease are observed

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L. Siu, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Quintela-Fandino M, Le Tourneau C, Duran I, Chen EX, Wang L, Tsao M, Bandarchi-Chamkhaleh B, Pham NA, Do T, MacLean M, Nayyar R, Tusche MW, Metser U, Wright JJ, Mak TW, Siu LL. Phase I combination of sorafenib and erlotinib therapy in solid tumors: safety, pharmacokinetic, and pharmacodynamic evaluation from an expansion cohort. Mol Cancer Ther. 2010 Mar;9(3):751-60. doi: 10.1158/1535-7163.MCT-09-0868. Epub 2010 Mar 2. PMID 20197396
- [Result] Duran I, Hotte SJ, Hirte H, Chen EX, MacLean M, Turner S, Duan L, Pond GR, Lathia C, Walsh S, Wright JJ, Dancey J, Siu LL. Phase I targeted combination trial of sorafenib and erlotinib in patients with advanced solid tumors. Clin Cancer Res. 2007 Aug 15;13(16):4849-57. doi: 10.1158/1078-0432.CCR-07-0382. PMID 17699864